CLINICAL TRIAL: NCT03104712
Title: The Importance of Glycemic Index on Postprandial Glycemia and Insulinemia in the Context of the Addition of Fat to Carbohydrate Foods: A Randomized Controlled Trial on Spaghetti Versus Rice as Mixed Meals
Brief Title: A Trial on the GI of Spaghetti Versus Rice as Mixed Meals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Parma (Other)
Responsible Party: Principal Investigator, Francesca Scazzina Ph.D., Assistant Professor, University of Parma
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Pasta+Sauces
Record Dates: First submitted 2017-03-27; First posted 2017-04-07 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Dietary Modification
Keywords: glycemic index
MeSH Terms: interventions — Glucose

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be unaware of the intervention associated with the samples being analyzed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Glucose #1 (Other): 50 grams of available carbohydrate from glucose monohydrate will be dissolved in 250mL water and consumed as a test meal
  Interventions: Other: Glucose #1
- Spaghetti (Active Comparator): 50 grams of available carbohydrate from spaghetti will be cooked according to package instructions and consumed as a test meal
  Interventions: Other: Spaghetti
- Rice (Active Comparator): 50 grams of available carbohydrate from white rice will be cooked according to package instructions and consumed as a test meal
  Interventions: Other: Rice
- Spaghetti + tomato sauce (Active Comparator): 50 grams of available carbohydrate from spaghetti plus tomato sauce (1:1 ratio) will be cooked according to package instructions and consumed as a test meal
  Interventions: Other: Spaghetti + Tomato Sauce
- Rice + tomato sauce (Active Comparator): 50 grams of available carbohydrate from white rice plus tomato sauce (1:1 ratio) will be cooked according to package instructions and consumed as a test meal
  Interventions: Other: Rice + Tomato Sauce
- Spaghetti + Pesto (Active Comparator): 50 grams of available carbohydrate from spaghetti plus pesto sauce (1:0.5 ratio) will be cooked according to package instructions and consumed as a test meal
  Interventions: Other: Spaghetti + Pesto
- Rice + Pesto (Active Comparator): 50 grams of available carbohydrate from white rice plus pesto sauce (1:0.5 ratio) will be cooked according to package instructions and consumed as a test meal
  Interventions: Other: Rice + Pesto
- Glucose #2 (Other): 50 grams of available carbohydrate from glucose monohydrate will be dissolved in 250mL water and consumed as a test meal
  Interventions: Other: Glucose #2
- Glucose #3 (Other): 50 grams of available carbohydrate from glucose monohydrate will be dissolved in 250mL water and consumed as a test meal
  Interventions: Other: Glucose #3

INTERVENTIONS:
Other: Glucose #1 — 50g available carbohydrate
  Other Names: Glucose Monohydrate
  Arms: Glucose #1
Other: Glucose #2 — 50g available carbohydrate
  Other Names: Glucose Monohydrate
  Arms: Glucose #2
Other: Glucose #3 — 50g available carbohydrate
  Other Names: Glucose Monohydrate
  Arms: Glucose #3
Other: Spaghetti — 50g available carbohydrate
  Arms: Spaghetti
Other: Rice — 50g available carbohydrate
  Other Names: white rice
  Arms: Rice
Other: Spaghetti + Tomato Sauce — 50g available carbohydrate
  Arms: Spaghetti + tomato sauce
Other: Rice + Tomato Sauce — 50g available carbohydrate
  Other Names: white rice + tomato sauce
  Arms: Rice + tomato sauce
Other: Spaghetti + Pesto — 50g available carbohydrate
  Arms: Spaghetti + Pesto
Other: Rice + Pesto — 50g available carbohydrate
  Other Names: white rice + pesto
  Arms: Rice + Pesto

SUMMARY:
Pasta and rice are two of the most commonly consumed grains worldwide, where the former has a low GI (e.g. spaghetti) and the latter, usually (as it depends on the type) has a higher GI (e.g. white rice). The most typical ways in which pasta and rice are consumed are with the addition of oil or tomato sauce, and are recommended to be consumed in this way in the Mediterranean diet. The Mediterranean diet has been demonstrated to reduce the risk of cardiovascular disease, improve glycemic control and is encouraged in many clinical guidelines globally for both cardiovascular risk reduction. Some studies have explored the differences in glycemic response of different carbohydrate foods consumed with the addition of fat demonstrating that the glycemic response is indeed reduced.However, the GI may remain of importance even when other means to reduce glycemic response are introduced.

The investigators therefore designed a randomized controlled crossover study to explore whether the addition of fat in the form of commonly consumed sauces which are recommended as part of a Mediterranean diet, affects the difference in glycemic response between a commonly consumed low GI and a higher GI carbohydrate food.

DETAILED DESCRIPTION:
Background:

Pasta and rice are two of the most commonly consumed grains worldwide, where the former has a low GI (e.g. spaghetti) and the latter, usually (as it depends on the type) has a higher GI (e.g. white rice). Low GI foods have been demonstrated to improve glycemic control, insulin sensitivity and diabetes management, and have been associated with reduced risk of chronic disease, including coronary heart disease. Therefore, GI is of importance as a potential dietary strategy to reduce postprandial glycemia and improve glycemic control, particularly with the increasing rates of diabetes.

Several studies have demonstrated how the addition of fat to a meal can reduce the glycemic response, some of which have suggested in a dose response manner. The mechanism by which increasing fat reduces the glycemic response may be through the effects on gastric emptying. Fat may modulate the gut hormones cholecystokinin (CCK) and peptide YY, which delay gastric emptying, which is known to be a major determinant of postprandial glycemia where small changes can have a substantial effect. Low GI foods result in lower glycemic excursions compared to higher GI foods, which, in addition to gastric emptying, may exert this effect through various pathways. Thus, there is importance of exploring the potential additional benefit beyond reducing the glycemic response with the addition of fat.

The most typical ways in which pasta and rice are consumed are with the addition of oil or tomato sauce, and are recommended to be consumed in this way in the Mediterranean diet. Among many benefits, the Mediterranean diet has been demonstrated to reduce the risk of cardiovascular disease, improved glycemic control and is encouraged in many clinical guidelines globally for both cardiovascular risk reduction and for diabetes. Some studies have explored the differences in glycemic response of different carbohydrate foods consumed with the addition of fat demonstrating that the glycemic response is indeed reduced.However, the GI may remain of importance even when other means to reduce glycemic response are introduced.

The investigators therefore designed a randomized controlled crossover study to explore whether the addition of fat in the form of commonly consumed sauces which are recommended as part of a Mediterranean diet, affects the difference in glycemic response between a commonly consumed low GI and a higher GI carbohydrate food.

Objective:

To assess whether the addition of fat to a low GI and higher GI carbohydrate food lowers the glycemic response equivalently, thus whether the difference between the low and higher GI food is preserved.

Scope:

The principal scope of the study is to evaluate the impact of two carbohydrate-containing foods varying in glycemic index, spaghetti and rice, on postprandial glucose.

To confirm that the two foods vary in GI, the GI of the rice will first be tested in Part A, since the GI of spaghetti has already been determined in the investigator's lab.

In Part B of the study, following the consumption of the test foods by healthy volunteers (see Study Design), the investigators will evaluate the differences in postprandial glucose, as well as insulin and c-peptide.

Implications:

These results will determine whether there is an independent effect of the GI of a carbohydrate containing food when fat is added to a meal in the context of how is it commonly and recommended to be consumed. These results may be useful to encourage the use of low GI foods for greater improvements in glycemic and insulinemic control, which is an important public health concern in today's global society.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy

Exclusion Criteria:

* BMI≥30kg/m2
* have any health conditions (including anemia and metabolic conditions such as hypertension, dyslipidemia, impaired glucose intolerance or diabetes)
* have celiac disease
* perform intense physical activity (LAF ≥2.10 - LARN 2014)
* currently taking any prescription medication for chronic diseases (including psychiatric)
* dietary supplements affecting the metabolism
* Women who are pregnant or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2018-03-12 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Glycemic Index | 2 hours (-10 and 0 -fasting-, 15, 30, 45, 60, 90, 120 minutes)
  postprandial response for glucose (IAUC); Comparisons will be made between the spaghetti and rice IAUCs in each of the 3 contexts (alone, with tomato sauce, with pesto)

SECONDARY OUTCOMES:
Postprandial Insulin | 2 hours (-10 and 0 -fasting-, 15, 30, 45, 60, 90, 120 minutes)
  postprandial response for plasma insulin (IAUC)
Postprandial C-peptide | 2 hours (-10 and 0 -fasting-, 15, 30, 45, 60, 90, 120 minutes)
  postprandial response for plasma c-peptide (IAUC)
Peak Glucose | 2 hours (-10 and 0 -fasting-, 15, 30, 45, 60, 90, 120 minutes)
  maximum value of postprandial glucose response

OTHER OUTCOMES:
Satiety using a 100cm visual analog scale | 2 hours
  differences in subject-rated satiety using a 100cm visual analog scale
Palatability using a 100cm visual analog scale | 12 minutes
  differences in subject-rated palatability using a 100cm visual analog scale
Gastrointestinal Symptoms using a questionnaire | 2 hours
  differences in subject-rated gastrointestinal symptom questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Scazzina, PhD, Principal Investigator — Department of Food and Drug, University of Parma; Furio Brighenti, PhD, Study Director — Department of Food and Drug, University of Parma
Locations (1):
- Department of Food and Drug, University of Parma, Parma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ajala O, English P, Pinkney J. Systematic review and meta-analysis of different dietary approaches to the management of type 2 diabetes. Am J Clin Nutr. 2013 Mar;97(3):505-16. doi: 10.3945/ajcn.112.042457. Epub 2013 Jan 30. PMID 23364002
- [Background] Barclay AW, Petocz P, McMillan-Price J, Flood VM, Prvan T, Mitchell P, Brand-Miller JC. Glycemic index, glycemic load, and chronic disease risk--a meta-analysis of observational studies. Am J Clin Nutr. 2008 Mar;87(3):627-37. doi: 10.1093/ajcn/87.3.627. PMID 18326601
- [Background] Mirrahimi A, de Souza RJ, Chiavaroli L, Sievenpiper JL, Beyene J, Hanley AJ, Augustin LS, Kendall CW, Jenkins DJ. Associations of glycemic index and load with coronary heart disease events: a systematic review and meta-analysis of prospective cohorts. J Am Heart Assoc. 2012 Oct;1(5):e000752. doi: 10.1161/JAHA.112.000752. Epub 2012 Oct 25. PMID 23316283
- [Background] Moghaddam E, Vogt JA, Wolever TM. The effects of fat and protein on glycemic responses in nondiabetic humans vary with waist circumference, fasting plasma insulin, and dietary fiber intake. J Nutr. 2006 Oct;136(10):2506-11. doi: 10.1093/jn/136.10.2506. PMID 16988118
- [Background] Thomas D, Elliott EJ. Low glycaemic index, or low glycaemic load, diets for diabetes mellitus. Cochrane Database Syst Rev. 2009 Jan 21;2009(1):CD006296. doi: 10.1002/14651858.CD006296.pub2. PMID 19160276
- [Background] Pironi L, Stanghellini V, Miglioli M, Corinaldesi R, De Giorgio R, Ruggeri E, Tosetti C, Poggioli G, Morselli Labate AM, Monetti N, et al. Fat-induced ileal brake in humans: a dose-dependent phenomenon correlated to the plasma levels of peptide YY. Gastroenterology. 1993 Sep;105(3):733-9. doi: 10.1016/0016-5085(93)90890-o. PMID 8359644
- [Background] Moran TH, Kinzig KP. Gastrointestinal satiety signals II. Cholecystokinin. Am J Physiol Gastrointest Liver Physiol. 2004 Feb;286(2):G183-8. doi: 10.1152/ajpgi.00434.2003. PMID 14715515
- [Background] Horowitz M, Edelbroek MA, Wishart JM, Straathof JW. Relationship between oral glucose tolerance and gastric emptying in normal healthy subjects. Diabetologia. 1993 Sep;36(9):857-62. doi: 10.1007/BF00400362. PMID 8405758
- [Background] Rayner CK, Samsom M, Jones KL, Horowitz M. Relationships of upper gastrointestinal motor and sensory function with glycemic control. Diabetes Care. 2001 Feb;24(2):371-81. doi: 10.2337/diacare.24.2.371. PMID 11213895
- [Background] Estruch R, Ros E, Salas-Salvado J, Covas MI, Corella D, Aros F, Gomez-Gracia E, Ruiz-Gutierrez V, Fiol M, Lapetra J, Lamuela-Raventos RM, Serra-Majem L, Pinto X, Basora J, Munoz MA, Sorli JV, Martinez JA, Martinez-Gonzalez MA; PREDIMED Study Investigators. Primary prevention of cardiovascular disease with a Mediterranean diet. N Engl J Med. 2013 Apr 4;368(14):1279-90. doi: 10.1056/NEJMoa1200303. Epub 2013 Feb 25. PMID 23432189 (Retraction: PMID 29897867 N Engl J Med. 2018 Jun 21;378(25):2441-2442)
- [Background] Esposito K, Maiorino MI, Bellastella G, Chiodini P, Panagiotakos D, Giugliano D. A journey into a Mediterranean diet and type 2 diabetes: a systematic review with meta-analyses. BMJ Open. 2015 Aug 10;5(8):e008222. doi: 10.1136/bmjopen-2015-008222. PMID 26260349
- [Background] Anderson TJ, Gregoire J, Pearson GJ, Barry AR, Couture P, Dawes M, Francis GA, Genest J Jr, Grover S, Gupta M, Hegele RA, Lau DC, Leiter LA, Lonn E, Mancini GB, McPherson R, Ngui D, Poirier P, Sievenpiper JL, Stone JA, Thanassoulis G, Ward R. 2016 Canadian Cardiovascular Society Guidelines for the Management of Dyslipidemia for the Prevention of Cardiovascular Disease in the Adult. Can J Cardiol. 2016 Nov;32(11):1263-1282. doi: 10.1016/j.cjca.2016.07.510. Epub 2016 Jul 25. PMID 27712954
- [Background] Canadian Diabetes Association Clinical Practice Guidelines Expert Committee; Dworatzek PD, Arcudi K, Gougeon R, Husein N, Sievenpiper JL, Williams SL. Nutrition therapy. Can J Diabetes. 2013 Apr;37 Suppl 1:S45-55. doi: 10.1016/j.jcjd.2013.01.019. Epub 2013 Mar 26. No abstract available. PMID 24070963
- [Background] Evert AB, Boucher JL, Cypress M, Dunbar SA, Franz MJ, Mayer-Davis EJ, Neumiller JJ, Nwankwo R, Verdi CL, Urbanski P, Yancy WS Jr; American Diabetes Association. Nutrition therapy recommendations for the management of adults with diabetes. Diabetes Care. 2013 Nov;36(11):3821-42. doi: 10.2337/dc13-2042. Epub 2013 Oct 9. PMID 24107659
- [Background] American Diabetes Association. (4) Foundations of care: education, nutrition, physical activity, smoking cessation, psychosocial care, and immunization. Diabetes Care. 2015 Jan;38 Suppl:S20-30. doi: 10.2337/dc15-S007. No abstract available. PMID 25537702
- [Background] Vinoy S, Lesdéma A, Cesbron-Lavau G, Goux A, and Meynier A. Chapter 13 Creating Food Products with a Lower Glycemic Index. The Glycemic Index: Applications in Practice. Taylor & Francis Group, 6000 Broken Sound Parkway NW, Suite 300, Boca Raton, FL 33487-2742 CRC Press. Pages 285-318.
- [Derived] Chiavaroli L, Di Pede G, Dall'Asta M, Cossu M, Francinelli V, Goldoni M, Scazzina F, Brighenti F. The importance of glycemic index on post-prandial glycaemia in the context of mixed meals: A randomized controlled trial on pasta and rice. Nutr Metab Cardiovasc Dis. 2021 Feb 8;31(2):615-625. doi: 10.1016/j.numecd.2020.09.025. Epub 2020 Sep 28. PMID 33229200